CLINICAL TRIAL: NCT01008956
Title: Immunogenicity and Safety Study of GSK Biologicals' Pandemic Influenza (H1N1) Candidate Vaccine GSK2340274A in Adults 18 to 64 Years of Age
Brief Title: Safety and Immune Response of One-Dose of Candidate H1N1 Influenza Vaccine GSK2340274A in Adults
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was cancelled before enrolment for reasons not related to vaccine safety or efficacy.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113924
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Influenza
Keywords: Influenza; H1N1; Pandemic; GSK Bio's influenza vaccine GSK2340274A
MeSH Terms: conditions — Influenza, Human

ARMS (1):
- Single Group (Experimental): Subjects enrolled in this group will be stratified by age (18 to 40 years and 41 to 64 years)
  Interventions: Biological: GSK Biologicals' investigational H1N1 Influenza Vaccine - GSK2340274A

INTERVENTIONS:
Biological: GSK Biologicals' investigational H1N1 Influenza Vaccine - GSK2340274A — Intramuscular injection, one dose

SUMMARY:
This study is designed to characterize the safety and immunogenicity of a' pandemic influenza (H1N1) candidate vaccine GSK2340274A in adults 18 to 64 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Indian male or female adults 18 to 64 years of age at time of the first vaccination, inclusive.
* Written informed consent obtained from the subject
* Good general health as assessed by medical history and physical examination.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line or mobile, but NOT a pay phone or other multiple-user device (i.e., a common-use phone serving multiple rooms or apartments)
* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:
* has practiced adequate contraception for 30 days prior to vaccination, and
* has a negative pregnancy test on the day of vaccination, and
* has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Medical history of physician-confirmed infection with an A/California/7/2009 (H1N1)v-like virus.
* Previous vaccination at any time with an A/California/7/2009 (H1N1)v-like virus vaccine.
* Presence or evidence of substance abuse or of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence of a temperature >= 38.0ºC (>=100.4ºF) by any route or method, or acute symptoms greater than "mild" severity on the scheduled date of first vaccination. NOTE: The subject may be vaccinated at a later date, provided symptoms have resolved, vaccination occurs within the window specified by the protocol, and all other eligibility criteria continue to be satisfied.
* Presence of significant acute or chronic, uncontrolled medical or psychiatric illness ("uncontrolled" is defined as requiring institution of new medical or surgical treatment or a significant alteration in the dose of an ongoing medication for uncontrolled symptoms, illness manifestations or drug toxicity within 3 months preceding the receipt of study vaccine).
* Diagnosed with cancer, or treatment for cancer within 3 years.
* Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible.
* Persons with a history of histologically-confirmed basal cell carcinoma of the skin successfully treated with local excision only are accepted and may enrol, but other histologic types of skin cancer are exclusionary.
* Women who are disease-free 3 years or more after treatment for breast cancer and receiving long-term prophylactic tamoxifen are excepted and may enrol.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination (no laboratory testing required).
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune modifying drugs within 6 months of study enrolment or planned administration during the study period. For corticosteroids, this will mean a dose equivalent to 10 mg/day of prednisone or equivalent when administered for > 2 weeks. Topical, intra-articular or inhaled and topical steroids are allowed.
* Receipt of any immunoglobulins and/or any blood products within 3 months of study enrolment or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin outside of 24 hours prior to vaccination are eligible. Persons receiving prophylactic antiplatelet medications, e.g., low-dose aspirin, and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome within 6 weeks of receipt of seasonal influenza vaccine.
* With the exception of seasonal influenza vaccination, administration of any vaccines within 30 days before vaccination. Seasonal influenza vaccine may be administered up to 14 days prior to study vaccination.
* Planned administration of any vaccine not foreseen by the study protocol from vaccination up to blood sampling at Day 21 including seasonal influenza vaccine or a monovalent pandemic H1N1 vaccine other than the study vaccine.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the receipt of study vaccine, or planned use during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines or component used in the manufacturing process of the study vaccine; a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Known pregnancy or a positive urine beta-human chorionic gonadotropin (ß-hCG) test result prior to the time of vaccination.
* Lactating or nursing female.
* Any conditions which, in the opinion of the investigator, prevents the subjects from participating in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Humoral immune response in terms of Hemagglutination Inhibition (HI) antibodies (Vaccine virus-homologous responses) | At Day 21 after vaccination

SECONDARY OUTCOMES:
Humoral immune response in terms of HI antibodies against A/California/7/2009 (H1N1)v-like antigen and any drifted strains | At Day 0, 21 and 182 after vaccination
Humoral immune response in terms of neutralizing antibodies against A/California/7/2009 (H1N1)v-like antigen and any drifted strains | At Day 0, 21 and 182 after vaccination
Occurrence of solicited local and general symptoms | During a 7-day (Day 0-6) follow-up period after vaccination.
Occurrence of unsolicited adverse events | During a 21-day (Day 0-20) follow-up period after vaccination and from Days 0 to 84.
Occurrence of medically attended and/or serious adverse events, and of potentially immune-mediated diseases. | From the beginning up to the end of the study (Day 182)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline